CLINICAL TRIAL: NCT00163826
Title: Optimisation of Patient Management Through Expediting the Spinal Clearance Process in the Major Trauma Patient
Brief Title: Spinal Clearance Study: Expediting the Spinal Clearance Process in the Major Trauma Patient
Status: Completed | Type: Observational
Sponsor: Bayside Health (Other Government)
Collaborators: Victorian Trauma Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 163/03
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Trauma; Traumatic Brain Injury; Spinal Injuries
Keywords: cervical spine injury; multiple trauma
MeSH Terms: conditions — Multiple Trauma; Brain Injuries, Traumatic; Spinal Injuries

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trauma Patients: Major trauma patients

SUMMARY:
The Alfred Hospital receives approximately 40% of the major trauma patients in Victoria, all of whom are at risk for spinal injuries. The potential for spinal injuries necessitates the undertaking of appropriate spinal investigations, and a delay in the completion of these investigations exposes the patient to the risk of a missed diagnosis of spinal instability and of complications of immobility; the potential spinal patient is required to wear a neck collar and be nursed lying flat whilst awaiting the completion and the appropriate documentation of spinal X-ray investigations.

The purpose of this study is to identify the issues causing a delay in the process of the completion of the appropriate spinal investigations and the documentation of the results.

The outcome of the proposed research will be the development of a clinical management protocol to expedite the process, with the aim of optimising patient care and reducing complications.

ELIGIBILITY:
Inclusion Criteria:

* Major trauma patients

Exclusion Criteria:

* Patients not subjected to spinal position restrictions on admission
* Patients deceased prior to spinal clearance
* Patients transferred to another centre prior to spinal clearance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital trauma patients
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2004-03; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen M Ackland, MHSc, Principal Investigator — Bayside Health
Locations (1):
- Bayside Health, Melbourne, Victoria, Australia